CLINICAL TRIAL: NCT01792518
Title: A Phase IIIb, Multicenter, Multinational, Randomized, Double-blind, Placebo Controlled, Parallel Group Study to Evaluate the Glycemic and Renal Efficacy of Once Daily Administration of Linagliptin 5 mg for 24 Weeks in Type 2 Diabetes Patients, With Micro- or Macroalbuminuria (30-3000mg/g Creatinine) on Top of Current Treatment With Angiotensin ConvEnzyme Inhibitor or Angiotensin Receptor Blocker - MARLINA (Efficacy, Safety & Modification of Albuminuria in Type 2 Diabetes Subjects With Renal Disease With LINAgliptin)
Brief Title: MARLINA - T2D : Efficacy, Safety & Modification of Albuminuria in Type 2 Diabetes Subjects With Renal Disease With LINAgliptin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.89; 2012-002603-17 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (2):
- linagliptin 5mg (Experimental): linagliptin 5 mg once daily
  Interventions: Drug: Linagliptin 5mg
- placebo (Placebo Comparator): matching placebo for linagliptin dose once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Arms: placebo
Drug: Linagliptin 5mg
  Arms: linagliptin 5mg

SUMMARY:
Evaluate linagliptin in terms of glycemic control as defined by HbA1c after 24 weeks of treatment and in terms of renal efficacy as defined by changes in albuminuria (UACR) after 24 weeks of treatment.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of type 2 diabetes mellitus
* Glycosylated Hemoglobin (HbA1c) between 6.5 and 10% (inclusive)
* Current therapy with ACEi or ARB at stable dose for 10 weeks
* Urinary albumin-to-creatinine ratio (UACR): 30-3000 mg/g creatinine documented in the previous 12 months or detected at Screening.
* Estimated Glomerular Filtration Rate (eGFR) greater than 30 ml/min.
* Age between 18 and 80 years.

Exclusion criteria:

* Dual or triple blockade of the Renin Angiotensin System (RAS)
* Uncontrolled hyperglycaemia
* Mean arterial blood pressure > 110 mmHg
* Known hypersensitivity or allergy to the investigational product, or their excipients (including matching placebos).
* Treatment with a glitazone within 6 months prior to informed consent.
* Treatment with a DiPeptidyl-Peptidase 4 (DPP-4) inhibitor, a Glucagon Like Peptide-1 (GLP-1) agonist, a Sodium/Glucose coTransporter 2 (SGLT2) inhibitor, a dopamine-agonist, a bile-acid sequestrant a short acting (prandial) insulin or premixed insulin within 10 weeks prior to informed consent.
* Treatment with anti-obesity drugs 10 weeks prior to informed consent.
* Alcohol or drug abuse within 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures or study drug intake in the opinion of the investigator.
* Current treatment with systemic steroids (glucocorticoids) at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent.
* Participation in another trial with an investigational drug within 2 months prior to informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2013-02; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (74):
- United States (15):
  - Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - Boehringer Ingelheim Investigational Site, Long Beach, California
  - Boehringer Ingelheim Investigational Site, North Hollywood, California
  - Boehringer Ingelheim Investigational Site, Denver, Colorado
  - Boehringer Ingelheim Investigational Site, Miami, Florida
  - Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - Boehringer Ingelheim Investigational Site, Flint, Michigan
  - Boehringer Ingelheim Investigational Site, Jackson, Mississippi
  - Boehringer Ingelheim Investigational Site, Asheboro, North Carolina
  - Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - Boehringer Ingelheim Investigational Site, Fargo, North Dakota
  - Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - Boehringer Ingelheim Investigational Site, Knoxville, Tennessee
  - Boehringer Ingelheim Investigational Site, Houston, Texas
- Canada (8):
  - Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - Boehringer Ingelheim Investigational Site, Mount Pearl, Newfoundland and Labrador
  - Boehringer Ingelheim Investigational Site, London, Ontario
  - Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - Boehringer Ingelheim Investigational Site, Waterloo, Ontario
- Denmark (4):
  - Boehringer Ingelheim Investigational Site, Gentofte Municipality
  - Boehringer Ingelheim Investigational Site, Hillerød
  - Boehringer Ingelheim Investigational Site, Silkeborg
  - Boehringer Ingelheim Investigational Site, Slagelse
- Finland (4):
  - Boehringer Ingelheim Investigational Site, Kerava
  - Boehringer Ingelheim Investigational Site, Oulu
  - Boehringer Ingelheim Investigational Site, Tampere
  - Boehringer Ingelheim Investigational Site, Turku
- France (8):
  - Boehringer Ingelheim Investigational Site, Bersée
  - Boehringer Ingelheim Investigational Site, Bourg-des-Comptes
  - Boehringer Ingelheim Investigational Site, Grenoble
  - Boehringer Ingelheim Investigational Site, Le Creusot
  - Boehringer Ingelheim Investigational Site, Marseille
  - Boehringer Ingelheim Investigational Site, Saint-Mandé
  - Boehringer Ingelheim Investigational Site, Vénissieux
  - Boehringer Ingelheim Investigational Site, Vieux-Condé
- Germany (7):
  - Boehringer Ingelheim Investigational Site, Aschaffenburg
  - Boehringer Ingelheim Investigational Site, Aßlar
  - Boehringer Ingelheim Investigational Site, Dresden
  - Boehringer Ingelheim Investigational Site, Düsseldorf
  - Boehringer Ingelheim Investigational Site, Flörsheim
  - Boehringer Ingelheim Investigational Site, Pirna
  - Boehringer Ingelheim Investigational Site, Schweinfurt
- Japan (7):
  - Boehringer Ingelheim Investigational Site, Aoba-ku,Sendai,Miyagi
  - Boehringer Ingelheim Investigational Site, Chiyoda-ku,Tokyo
  - Boehringer Ingelheim Investigational Site, Cyuo-ku,Tokyo
  - Boehringer Ingelheim Investigational Site, Kita-ku, Osaka, Osaka
  - Boehringer Ingelheim Investigational Site, Shimizu-ku,Shizuoka city,Shizuoka
  - Boehringer Ingelheim Investigational Site, Suita,Osaka
  - Boehringer Ingelheim Investigational Site, Teine-ku,Sapporo,Hokkaido
- Philippines (3):
  - Boehringer Ingelheim Investigational Site, Cebu City, Philippines
  - Boehringer Ingelheim Investigational Site, Pasig City, Philippines
  - Boehringer Ingelheim Investigational Site, San Juan City, Philippines
- South Korea (5):
  - Boehringer Ingelheim Investigational Site, Goyang
  - Boehringer Ingelheim Investigational Site, Jinju
  - Boehringer Ingelheim Investigational Site, Seongnam
  - Boehringer Ingelheim Investigational Site, Seoul
  - Boehringer Ingelheim Investigational Site, Wŏnju
- Spain (5):
  - Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - Boehringer Ingelheim Investigational Site, Madrid
  - Boehringer Ingelheim Investigational Site, Pozuelo de Alarcón
  - Boehringer Ingelheim Investigational Site, San Sebastián de los Reyes
  - Boehringer Ingelheim Investigational Site, Valencia
- Taiwan (6):
  - Boehringer Ingelheim Investigational Site, Changhua
  - Boehringer Ingelheim Investigational Site, Kaohsiung City
  - Boehringer Ingelheim Investigational Site, New Taipei City
  - Boehringer Ingelheim Investigational Site, Taichung
  - Boehringer Ingelheim Investigational Site, Tainan
  - Boehringer Ingelheim Investigational Site, Taipei
- Vietnam (2):
  - Boehringer Ingelheim Investigational Site, Hanoi, Vietnam
  - Boehringer Ingelheim Investigational Site, Ho Chi Minh City

REFERENCES:
- [Derived] Siwy J, Klein T, Rosler M, von Eynatten M. Urinary Proteomics as a Tool to Identify Kidney Responders to Dipeptidyl Peptidase-4 Inhibition: A Hypothesis-Generating Analysis from the MARLINA-T2D Trial. Proteomics Clin Appl. 2019 Mar;13(2):e1800144. doi: 10.1002/prca.201800144. Epub 2019 Jan 28. PMID 30632692
- [Derived] Groop PH, Cooper ME, Perkovic V, Hocher B, Kanasaki K, Haneda M, Schernthaner G, Sharma K, Stanton RC, Toto R, Cescutti J, Gordat M, Meinicke T, Koitka-Weber A, Thiemann S, von Eynatten M. Linagliptin and its effects on hyperglycaemia and albuminuria in patients with type 2 diabetes and renal dysfunction: the randomized MARLINA-T2D trial. Diabetes Obes Metab. 2017 Nov;19(11):1610-1619. doi: 10.1111/dom.13041. Epub 2017 Jul 31. PMID 28636754
- [Derived] Groop PH, Cooper ME, Perkovic V, Sharma K, Schernthaner G, Haneda M, Hocher B, Gordat M, Cescutti J, Woerle HJ, von Eynatten M. Dipeptidyl peptidase-4 inhibition with linagliptin and effects on hyperglycaemia and albuminuria in patients with type 2 diabetes and renal dysfunction: Rationale and design of the MARLINA-T2D trial. Diab Vasc Dis Res. 2015 Nov;12(6):455-62. doi: 10.1177/1479164115579002. Epub 2015 Jul 28. PMID 26224765

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 360 patients were randomised and treated (Placebo: 178 patients, Linagliptin: 182 patients.)
Pre-assignment Details: Randomized, double-blind, placebo controlled, parallel group study to evaluate glycemic and renal efficacy of once daily administration of Linagliptin 5 milligram (mg) for 24 weeks in type 2 diabetes patients, with micro- or macroalbuminuria on top of current treatment with Angiotensin Converting Enzyme inhibitor or Angiotensin Receptor Blocker
Groups:
- Placebo: Patients received 1 matching placebo tablet to Linagliptin 5 mg, administered orally, once every day for 24 weeks during the double blind treatment period.
- Linagliptin 5 mg: Patients received 1 tablet of Linagliptin 5 mg, administered orally, once every day for 24 weeks during the double blind treatment period.
Period: Overall Study
Arm/Group | Placebo | Linagliptin 5 mg
Started | 178 | 182
Completed | 170 | 175
Not Completed | 8 | 7
Not completed — Adverse Event | 3 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Other Reason | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) - including all patients treated with at least one dose of randomised trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linagliptin 5 mg | Total
Number analyzed (Participants) | 178 | 182 | 360
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (9.3) | 61.0 (10.0) | 60.6 (9.6)
Gender [Count of Participants; unit: Participants]
  Female | 65 | 66 | 131
  Male | 113 | 116 | 229

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline After 24 Weeks Double-blind Randomized Treatment
Description: Change from baseline in Glycated haemoglobin (HbA1c) [%] after 24 weeks of treatment with double- blind trial medication. The term "baseline" refers to the last observation before the start of any randomised trial treatment. The number of participants analysed displays the number of participants with available data at the timepoint of interest.
Time Frame: Baseline and 24 weeks
Population: Full Analysis Set (FAS) - including all randomised patients who were treated with at least one dose of study drug, had a baseline HbA1c and a baseline Urinary albumin creatinine ratio (UACR), and at least one on treatment HbA1c or UACR assessment. Observed Case (OC): Values after the use of rescue medication were set to missing.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 156 | 161
Percentage of HbA1c | -0.03 (0.06) | -0.63 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Superiority of Linagliptin 5 mg vs. placebo: change in HbA1c is analysed using mixed model repeated measures (MMRM) approach. Model includes baseline HbA1c, baseline log10 (UACR), baseline HbA1c by visit and baseline log10 (UACR) by visit as linear covariates and treatment, visit, visit by treatment interaction as fixed effects; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The Unstructured covariance structure has been used to fit the mixed model; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-0.78 to -0.43], Standard Error of Mean 0.09 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as Linagliptin 5 mg minus Placebo

2. Secondary Outcome: The Time Weighted Average of Percentage Change From Baseline in UACR During the Course of 24 Weeks of Treatment
Description: The time weighted average of percentage change from baseline in UACR (mg/g creatinine) during the course of 24 weeks of treatment. The term "baseline" for UACR refers to the geometric mean of UACR values measured at Visits 2 and 3. The number of participants analysed displays the number of participants with available data at the timepoint of interest. The Least Squares Means are adjusted geometric means.
Time Frame: Baseline and 24 weeks
Population: Full Analysis Set (FAS) - including all randomised patients who were treated with at least one dose of study drug, had a baseline HbA1c and a baseline Urinary albumin creatinine ratio (UACR), and at least one on treatment HbA1c or UACR assessment. Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/g creatinine
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 173 | 178
mg/g creatinine | 0.9487 (0.06) [0.8857 to 1.0162] | 0.8902 (0.06) [0.8318 to 0.9526]
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Superiority of Linagliptin 5 mg vs. placebo: change in UACR is analysed using analysis of covariance model. Model includes baseline HbA1c and baseline log10 (UACR) as linear covariates and treatment as fixed effect; Test type: Superiority or Other; p = 0.1954, ANCOVA; Ratio of adjusted geometric means = 0.94, 95% CI 2-sided [0.85 to 1.03] — Ratio of relative change for Linagliptin 5 mg over placebo is presented

3. Secondary Outcome: The Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) After 24 Weeks of Treatment
Description: The change from baseline in estimated glomerular filtration rate (eGFR) as assessed by chronic kidney disease epidemiology collaboration (CKD-EPI) equation (cystatin C) after 24 weeks of treatment. The term "baseline" refers to the last observation before the start of any randomised trial treatment. The number of participants analysed displays the number of participants with available data at the timepoint of interest. This outcome measure is a secondary safety endpoint.
Time Frame: Baseline and 24 weeks
Population: Treated Set
Measure: Least Squares Mean (Standard Error); unit: milliliter/minute/1.73 square metre
Arm/Group | Placebo | Linagliptin 5 mg
Number analyzed (Participants) | 156 | 162
milliliter/minute/1.73 square metre | -2.35 (1.92) | -4.98 (1.89)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5 mg; Change in eGFR is analysed using mixed model repeated measures (MMRM) approach. Model includes baseline HbA1c, baseline log10 (UACR), baseline eGFR, baseline HbA1c by visit, baseline log10 (UACR) by visit and baseline eGFR by visit as linear covariates and treatment, visit, visit by treatment interaction as fixed effects; Test type: Superiority or Other; p = 0.3306, Mixed Models Analysis; The Unstructured covariance structure has been used to fit the mixed model; Mean Difference (Final Values) = -2.63, 95% CI 2-sided [-7.95 to 2.68], Standard Error of Mean 2.70 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as Linagliptin 5 mg minus Placebo

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after the last drug administration, up to 240 days
Arm/Group | Placebo | Linagliptin 5 mg
Serious Adverse Events (participants affected / at risk) | 8/178 | 17/182
Other Adverse Events (participants affected / at risk) | 27/178 | 39/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=178) | Linagliptin 5 mg (N=182)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 2
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Arteriovenous graft site infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Peripheral nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aortic occlusion (Vascular disorders) | 1 | 0
Necrosis ischaemic (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=178) | Linagliptin 5 mg (N=182)
Nasopharyngitis (Infections and infestations) | 10 | 13
Upper respiratory tract infection (Infections and infestations) | 9 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 10 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.